CLINICAL TRIAL: NCT01807806
Title: Safety and Effectiveness Study: Interactive Game-Based System for Psychological Health Education
Brief Title: Safety and Effectiveness Study: Role Playing Game for Friends and Family of Service Members
Acronym: RPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Soar Technology (Unknown); Creative Media and Behavioral Health Center (Unknown); USC Center for Innovation and Research on Veterans & Military Families (Other)
Responsible Party: Principal Investigator, Maryalice Jordan-Marsh, Associate professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: USC Subcontract No 10150.003.0
Record Dates: First submitted 2013-03-05; First posted 2013-03-08 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Communication
Keywords: veterans, military, families
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Role-playing game (Experimental): All eligible participants were invited to play the role playing game
  Interventions: Behavioral: Role-playing game

INTERVENTIONS:
Behavioral: Role-playing game — Eligible participants will be invited to engage with a role-playing game for 30 minutes. The role play presents situations where a service member/veteran interacts with family or friends.

SUMMARY:
This project is a partnership between Soar Technology, the University of Southern California (USC) Center for Innovation and Research on Veterans and Military Families (CIR) and the USC Creative Media and Behavioral Health Center (CM&BHC) to conduct a Safety and Effectiveness Study (SES) for an educational role-playing game developed by Soar Technology, Inc. The purpose of the intervention to be delivered by Soar Technology is to educate families and friends with the ultimate goal of empowering them to have a conversation with the veteran/service member about readjustment issues. The study will assess the safety and effectiveness of the provided game using personal interviews, play testing, and surveys. The game playing experience is hypothesized to be safe and effective with respect to having conversations with veterans/service members following deployment.

DETAILED DESCRIPTION:
The intervention is a multi-scenario role playing simulation. Participants view the scenario and answer questions about what has been displayed as typical for post deployment service members. Participants receive immediate feedback with respect to expectations set by simulation developers.

ELIGIBILITY:
Inclusion Criteria:

* must be friend or family member to a military veteran or service member who experienced a deployment no earlier than 2007, or who are currently active and have recently returned from a deployment
* be able to read English
* be reachable via cell phone
* age range 18-86
* daily access to the internet
* have a personal email account for contact
* experience with filling out online surveys, or online shopping, or social media, or playing digital games

Exclusion Criteria:

* no acute psychopathology based on PHQ-9 and VAS scores at baseline and VAS and PHQ-2 at pre-test
* must not be active duty military personnel or a veteran at the time of the study
* service member or self is not currently receiving treatment at VA or other mental health facility

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in mental health status at one week | One week
  Patient Health Questionnaire (PHQ) Depression Scale

SECONDARY OUTCOMES:
Change from intervention in task-based motivation at one week | Intervention, one week
  Intrinsic Motivation Inventory

OTHER OUTCOMES:
change from baseline to knowledge of best practices for post deployment conversations at one week | one week
  A knowledge acquisition inventory of strategies for approaching service members with post deployment readjustment issues
Change in anxiety from immediately after the intervention to rating one week later | one week
  visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Maryalice Jordan-Marsh, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California School of Social Work, Los Angeles, California, United States